CLINICAL TRIAL: NCT03101982
Title: Hyperbaric Oxygenation (HBO) in Traumatic Spinal Cord Injury. (EOS) - Pilot Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: less of patients enrolled
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBOwings
Record Dates: First submitted 2017-03-22; First posted 2017-04-05 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2023-03

CONDITIONS: Traumatic Injury of the Spinal Cord
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test (Active Comparator): HBO, ASIA score, blood taking
  Interventions: Drug: HBO
- control (No Intervention): ASIA score, blood taking

INTERVENTIONS:
Drug: HBO — Hyperbaric oxygenation (HBO) is defined as breathing of 100% oxygen under elevated ambient pressure in a hyperbaric chamber. HBO is considered a pharmacological therapy.
  Other Names: Hyperbaric oxygenation
  Arms: test

SUMMARY:
Hypothesis of the Study:

Based on the presented results, the investigator hypothesises that HBO preserves neurons that are not irreversibly damaged (i.e. severed) during initial trauma, thus enabling regain of their function. The investigator predicts that HBO treatment protects and enhances motor function in initially paralysed regions, including improvement in function of the extremities as well as recovery of urinary bladder control and bowel function.

Outline of the Proposed Study:

Within a prospective "proof of principle" trial, a total of 100 patients will be included. Fifty patients will be recruited at the Division of Thoracic and Hyperbaric Surgery, Medical University of Graz. In parallel, 50 control patients will be included at the Department of Orthopaedics and Trauma, Paracelsus University Salzburg, Salzburger Landeskliniken (SALK), Austria. Thereby, all patients that are admitted at the Medical University of Graz can be treated and the enrolment of 50 patients into the treatment group can be implemented within the outlined time frame. The active recruitment period is planned for three years. Both HBO treated and control patients will undergo the same surgical and nonsurgical procedures. HBO treatment will be started within 24 hours after the injury. A total of 21 consecutive daily sessions will be applied, followed by routine rehabilitation programmes. By matching control and HBO-treated patients, an evaluation of the treatment effect of HBO is possible. The outcome will be evaluated by implementing the American Spinal Injury Association (ASIA)-scores and magnet resonance (MR) imaging. Additionally, inflammatory and regenerative blood markers will be analysed (neuroendocrine markers/neuro-transmitters: S100beta, Brain Derived Neurotrophic Growth Factor [BDNF], Glial Fibrillary Acidic Protein [GFAP], Reactive Oxygen Species (ROS), norepinephrine; array of pro- and anti-inflammatory cytokines and chemokines).

ELIGIBILITY:
Inclusion Criteria:

Test cohort and control cohort:

* age: 16 to 70 years
* Traumatic spinal cord injury
* Initial incomplete or complete (ASIA) sensor/motoric dysfunction
* Mentally competent patient (no mental disability in history in case of intubated patient)
* No relevant neuromuscular diseases / neurological deficits before trauma
* Vertebral column stable, no relevant mechanical compression of spinal cord with our without surgical intervention within 24 hours after the injury;
* Spinal MRI and CT-scan within first 24 hours

Test cohort only:

* Cardiorespiratory situation allowing safe application of HBO
* Ability to equalize pressure differences in middle ear confirmed by an ENT (ear, nose, throat) physician or pretherapeutic myringotomy
* Circumstances allowing HBO-treatment to be started < 24 hours after the injury

Exclusion Criteria:

Test cohort and control cohort:

* Morphologically confirmed complete discontinuation of the spinal cord
* Cardio-respiratory instability
* Persistent seizure activity in spite of medication
* Craniocerebral injury exceeding mere commotion
* Pregnancy
* Sepsis, Systemic Inflammatory Response Syndrome (SIRS)
* Simultaneous participation in another interventional study if relevant

Test cohort only:

* Cystic or bullous lung disease, untreated pneumothorax
* Treatment with doxorubicin in patient´s history

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Improvement of neurological deficits caused by spinal cord lesions | Change from baseline-admission scores ( ASIA ) at 12 months
  assessed by American Spinal Injury Association (ASIA) scores
Correlation of clinical observations with blood parameters | Blood samples will be taken at the time of admission, immediately before the first HBO, immediately after the first HBO, on days 1, 3, 7, 14 , 21 before the respective HBO, and at the 35 days and two months follow-up
  assessed by routinely taken blood tests

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided